CLINICAL TRIAL: NCT02702180
Title: A Randomised, Double-blind, Placebo-controlled Multicentre Clinical Trial of Inhaled Molgramostim in Autoimmune Pulmonary Alveolar Proteinosis Patients
Brief Title: Efficacy and Safety of Inhaled Molgramostim (rhGM-CSF) in Autoimmune Pulmonary Alveolar Proteinosis
Acronym: IMPALA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Savara Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MOL-PAP-002; 2015-003878-33 (EudraCT Number)
Record Dates: First submitted 2016-02-28; First posted 2016-03-08 (Estimated); Results first posted 2022-04-15 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Autoimmune Pulmonary Alveolar Proteinosis
MeSH Terms: conditions — Pulmonary Alveolar Proteinosis, Acquired | interventions — molgramostim; regramostim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (4):
- Double-blind molgramostim once daily (Experimental): Inhalation of molgramostim nebuliser solution 300 mcg once daily for 24 weeks
  Interventions: Drug: Molgramostim; Device: PARI eFlow nebulizer system
- Double-blind molgramostim intermittent (Experimental): Inhalation of molgramostim nebuliser solution 300 mcg for 7 days and placebo nebuliser solution for 7 days for 24 weeks (12 cycles)
  Interventions: Drug: Molgramostim; Device: PARI eFlow nebulizer system
- Double-blind placebo (Placebo Comparator): Inhalation of placebo nebuliser solution once daily for 24 weeks
  Interventions: Drug: Placebo; Device: PARI eFlow nebulizer system
- Open-label molgramostim intermittent (Experimental): Inhalation of molgramostim nebuliser solution 300 mcg for 7 days and placebo nebuliser solution for 7 days for 24 or 48 weeks from completion of the double-blind period
  Interventions: Drug: Molgramostim; Device: PARI eFlow nebulizer system

INTERVENTIONS:
Drug: Molgramostim — 300 mcg molgramostim (rhGM-CSF) nebulizer solution for inhalation
  Other Names: rhGM-CSF
  Arms: Double-blind molgramostim intermittent; Double-blind molgramostim once daily; Open-label molgramostim intermittent
Drug: Placebo — Placebo nebulizer solution for inhalation
  Arms: Double-blind placebo
Device: PARI eFlow nebulizer system — PARI eFlow nebulizer system

SUMMARY:
This study evaluates inhaled molgramostim (recombinant human granulocyte macrophage-colony stimulating factor [rhGM-CSF]) in the treatment of autoimmune pulmonary alveolar proteinosis (aPAP) patients. A third of the patients will receive inhaled molgramostim once daily for 24 weeks, a third will receive inhaled molgramostim intermittently (7 days on, 7 days off) for 24 weeks and a third will receive inhaled matching placebo for 24 weeks.

DETAILED DESCRIPTION:
The trial is a phase 2, randomized, double-blind, placebo-controlled multicentre clinical trial investigating efficacy and safety of inhaled molgramostim (rhGM-CSF) in patients with aPAP.

The trial will include 2 periods; a double-blind treatment period consisting of up to 8 trial visits (Screening, Baseline, and at Weeks 4, 8,12, 16, 20 and 24 after randomisation) and a open-label follow-up period consisting of up to 5 trial visits (at Weeks 4, 12, 24, 36 and 48 post-treatment).

In the double-blind treatment period, eligible subjects will be randomised to treatment for up to 24 weeks with either: 1) inhaled molgramostim (300 µg) once daily (MOL-OD), 2) inhaled molgramostim (300 µg) and matching placebo administered intermittently (7 days on and 7 days off) (MOL-INT) or 3) inhaled placebo once daily (PBO). During the follow-up period, all participants will receive inhaled molgramostim intermittently (7 days on, 7 days off). During the trial, whole lung lavage (WLL) may be applied as rescue therapy in case of significant clinical worsening.

ELIGIBILITY:
Inclusion Criteria:

* aPAP diagnosed by computed tomography, or by biopsy, or by Broncho Alveolar Lavage (BAL), and by increased GM-CSF autoantibodies in serum.
* Stable or progressive aPAP during a minimum period of 2 months prior to the Baseline visit.
* Arterial oxygen tension (PaO2) <75 mmHg/<10 kilo Pascal (kPa) at rest, OR desaturation of >4 percentage points on the 6MWT
* An alveolar-arterial oxygen difference [(A-a)DO2] of minimum 25 mmHg/3.33 kPa
* Female or male ≥18 years of age
* Females who have been post-menopausal for >1 year or females of childbearing potential after a confirmed menstrual period using a highly efficient method of contraception (i.e. a method with <1% failure rate such as combined hormonal contraception, progesterone-only hormonal contraception, intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomised partner, sexual abstinence), during and until 30 days after last dose of double-blind trial treatment. Females of childbearing potential must have a negative serum pregnancy test at Screening (Visit 1) and a negative urine pregnancy test at dosing at Baseline (Visit 2) and must not be lactating
* Males agreeing to use condoms during and until 30 days after last dose of double-blind medication, or males having a female partner who is using adequate contraception as described above
* Willing and able to provide signed informed consent
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures specified in the protocol as judged by the investigator

Exclusion Criteria:

* Diagnosis of hereditary or secondary PAP
* WLL within 1 month of Baseline
* Treatment with GM-CSF within 3 months of Baseline
* Treatment with rituximab within 6 months of Baseline
* Treatment with plasmapheresis within 3 months of Baseline
* Treatment with any investigational medicinal product within 4 weeks of Screening
* Concomitant use of sputum modifying drugs such as carbocysteine or ambroxol
* History of allergic reactions to GM-CSF
* Connective tissue disease, inflammatory bowel disease or other autoimmune disorder requiring treatment associated with significant immunosuppression, e.g. more than 10 mg/day systemic prednisolone
* Previous experience of severe and unexplained side-effects during aerosol delivery of any kind of medicinal product
* History of, or present, myeloproliferative disease or leukaemia
* Known active infection (viral, bacterial, fungal or mycobacterial)
* Apparent pre-existing concurrent pulmonary fibrosis
* Any other serious medical condition which in the opinion of the investigator would make the participant unsuitable for the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2016-03-21 (Actual); Primary Completion 2019-04-19 (Actual); Study Completion 2019-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cliff Morgan, MD, Principal Investigator — Royal Brompton Hospital, London
Locations (30):
- United States (3):
  - UCLA, Los Angeles, California
  - University of Florida, Gainesville, Florida
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
- Royal Prince Alfred Hospital, Sydney, New South Wales, Australia
- Aarhus University Hospital, Aarhus, Denmark
- CHU Rennes Hospital Pontchaillou, Rennes, France
- Germany (4):
  - Westdeutsches Lungenzentrum am Universitätsklinikum Essen, Essen
  - Asklepios Fachkliniken München - Gauting, Gauting
  - Thoraxklinik am Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Schleswig-Holstein Zentralklinikum, Lübeck Medizinische Klinik III, Pneumologie, Lübeck
- Attikon University Hospital, Athens, Greece
- Rabin Medical Center, Petah Tikva, Israel
- IRCCS Policlinico San Matteo, Pavia, Italy
- Japan (5):
  - Niigata University Medical and Dental Hospital, Niigata
  - National Hospital Organization Kinki-Chuo, Osaka
  - Tohoku University Hospital, Sendai
  - Aichi Medical University Hospital, Toyohashi
  - Kanagawa Cardiovascular and Respiratory Center, Yokohama
- St. Antonius Hospital, Nieuwegein, Netherlands
- Portugal (2):
  - Hospital de dia de Pneumologia, Lisbon
  - Hospital Sao Joao, Porto
- City Hospital St. Petersburg, Saint Petersburg, Russia
- II. Pulmonary Department National Institut for TB, Lung Diseases and Chest Surgery, Vyšné Hágy, Slovakia
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Division of Pulmonary and Critical Care Medicine, Seoul
  - Samsung Medical Center, Division of Pulmonary and Critical Care Medicine, Seoul
- Hospital University de Bellvitge (HUB), Barcelona, Spain
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland
- Yedikule Pulmonary Diseases and Pulmonary Surgery Training and Research Hospital, Istanbul, Turkey (Türkiye)
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Trapnell BC, Inoue Y, Bonella F, Morgan C, Jouneau S, Bendstrup E, Campo I, Papiris SA, Yamaguchi E, Cetinkaya E, Ilkovich MM, Kramer MR, Veltkamp M, Kreuter M, Baba T, Ganslandt C, Tarnow I, Waterer G, Jouhikainen T; IMPALA Trial Investigators. Inhaled Molgramostim Therapy in Autoimmune Pulmonary Alveolar Proteinosis. N Engl J Med. 2020 Oct 22;383(17):1635-1644. doi: 10.1056/NEJMoa1913590. Epub 2020 Sep 7. PMID 32897035

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 30 sites in 18 countries (United Kingdom, Denmark, Germany, Italy, France, Greece, Switzerland, Spain, Portugal, Slovakia, Netherlands, Turkey, Russia, Israel, Japan, South Korea, Australia, and the US) enrolled participants in the trial. First participant was enrolled on 21 March 2016 and last subject completed the study on 27 September 2019.
Pre-assignment Details: A total of 235 participants were screened, and 138 were randomized and treated.
  1 participant in the MOL-INT group and 1 participant in the PBO group withdrew between the double-blind period and the open-label period. 1 participant who withdrew from the double-blind period entered the open-label period.
Groups:
- Molgramostim Once Daily: Inhalation of molgramostim nebuliser solution 300 mcg once daily for 24 weeks
  Molgramostim: 300 mcg molgramostim (rhGM-CSF) nebulizer solution for inhalation
  PARI eFlow nebulizer system: PARI eFlow nebulizer system
- Molgramostim Intermittent: Inhalation of molgramostim nebuliser solution 300 mcg for 7 days and placebo nebuliser solution for 7 days for 24 weeks (12 cycles)
  Molgramostim: 300 mcg molgramostim (rhGM-CSF) nebulizer solution for inhalation
  Placebo: Placebo nebulizer solution for inhalation
  PARI eFlow nebulizer system: PARI eFlow nebulizer system
- Placebo: Inhalation of placebo nebuliser solution once daily for 24 weeks
  Placebo: Placebo nebulizer solution for inhalation
  PARI eFlow nebulizer system: PARI eFlow nebulizer system
Period: Double-blind Treatment Period
Arm/Group | Molgramostim Once Daily | Molgramostim Intermittent | Placebo
Started | 46 | 45 | 47
Completed | 45 | 44 | 43
Not Completed | 1 | 1 | 4
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 2
Period: Open-label Treatment Period
Arm/Group | Molgramostim Once Daily | Molgramostim Intermittent | Placebo
Started | 45 | 43 | 43
Completed | 45 | 42 | 41
Not Completed | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Withdrawn in error | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Molgramostim Once Daily | Molgramostim Intermittent | Placebo | Total
Number analyzed (Participants) | 46 | 45 | 47 | 138
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 0 | 1
  Between 18 and 65 years | 34 | 37 | 41 | 112
  >=65 years | 12 | 7 | 6 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (13.32) | 49.2 (14.06) | 46.1 (14.84) | 49.8 (14.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 22 | 59
  Male | 28 | 26 | 25 | 79
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 25 | 13 | 11 | 49
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 20 | 32 | 36 | 88
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 0 | 4
  Japan | 20 | 10 | 10 | 40
  United Kingdom | 1 | 3 | 1 | 5
  Switzerland | 0 | 0 | 1 | 1
  Portugal | 0 | 1 | 2 | 3
  Russia | 1 | 1 | 6 | 8
  Spain | 0 | 1 | 1 | 2
  Greece | 1 | 0 | 3 | 4
  Netherlands | 2 | 3 | 1 | 6
  South Korea | 3 | 2 | 1 | 6
  Turkey | 4 | 4 | 2 | 10
  Denmark | 1 | 1 | 1 | 3
  Italy | 3 | 3 | 7 | 13
  Israel | 1 | 5 | 1 | 7
  Slovakia | 2 | 1 | 1 | 4
  France | 2 | 1 | 2 | 5
  Australia | 0 | 1 | 0 | 1
  Germany | 3 | 6 | 7 | 16
Smoking [Count of Participants; unit: Participants]
  Previous | 27 | 20 | 20 | 67
  Never | 13 | 16 | 16 | 45
  Current | 6 | 9 | 11 | 26
Time since aPAP diagnosis [Mean (Standard Deviation); unit: months] | 39.8 (58.12) | 40.0 (45.87) | 32.0 (31.50) | 37.2 (46.18)
Participants with previous whole lung lavage [Count of Participants; unit: Participants] | 23 | 31 | 30 | 84
Disease severity score (DSS) [Count of Participants; unit: Participants]
  DSS 1: No symptoms and PaO2 ≥70 mmHg | 4 | 5 | 3 | 12
  DSS 2: Symptomatic and PaO2 ≥70 mmHg | 12 | 14 | 16 | 42
  DSS 3: 60 mmHg ≤ PaO2 <70 mmHg | 17 | 13 | 14 | 44
  DSS 4: 50 mm Hg ≤ PaO2 <60 mmHg | 5 | 9 | 10 | 24
  DSS 5: PaO2 <50 mmHg | 8 | 4 | 4 | 16

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline of Alveolar-arterial Oxygen Concentration (A-a(DO2)) After 24 Weeks of Treatment
Description: Measurement of (A-a)DO2 was done by blood gas analysis. An arterial blood sample was collected in the supine position, after resting for at least 10 minutes (or longer if required to achieve stable oxygen saturation). The sample was analyzed for arterial oxygen tension (PaO2) and partial pressure of carbon dioxide (PaCO2). The calculation of (A-a)DO2 was done centrally by using a formula described in the protocol.
Time Frame: From baseline to 24 weeks
Population: Full analysis set (FAS): all randomized participants, analyzed according to randomized treatment. Not all participants in the FAS had blood gas analysis done at Week 24, therefore the overall number of participants analyzed is less than the total number of randomized participants.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Molgramostim Once Daily | Molgramostim Intermittent | Placebo
Number analyzed (Participants) | 45 | 43 | 43
mmHg | 28.6 (21.95) | 29.3 (17.96) | 32.0 (20.90)
Statistical Analysis 1: Comparison: Molgramostim Once Daily vs Placebo; Primary endpoint was evaluated using analysis of covariance with treatment, whole lung lavage within 2 months before baseline, and geographic region as factors, and baseline values as covariates. To control type I error, key secondary endpoints were analyzed using a testing hierarchy wherein once daily molgramostim and placebo was compared and if statistical significance was reached, evaluation of intermittent molgramostim and placebo would proceed; Test type: Superiority; p = 0.1688, ANCOVA; Least Square Means (LSmean) = -4.6, 95% CI 2-sided [-11.1 to 2.0] — The estimated value represents the estimated difference between once daily molgramostim and placebo groups in LSmean change from baseline to week 24
Statistical Analysis 2: Comparison: Molgramostim Intermittent vs Placebo; Test type: Superiority; p = 0.3968, ANCOVA; Least Square Means (LSmean) = -2.8, 95% CI 2-sided [-9.3 to 3.7] — The estimated value represents the estimated difference between intermittent molgramostim and placebo groups in LSmean change from baseline to week 24

2. Secondary Outcome: Change From Baseline in 6-minute Walking Distance (6MWD) After 24 Weeks of Treatment
Description: The 6MWD was assessed by the use of 6-minute walking test (6MWT). The 6MWT was performed in accordance with the 2014 ATS/ERS guideline "field walking tests in chronic respiratory disease" (Holland et al. 2014) by technicians with documented training and experience.
  Where possible, the test was conducted with the participant breathing ambient atmospheric air. If the participant required oxygen supplementation at rest, a titration procedure was carried out as part of the 6MWT at screening in order to determine the oxygen flow rate required for the participant to complete the test. This flow rate was to be used during subsequent tests, if possible.
Time Frame: From baseline to 24 weeks
Population: FAS. Not all participants in the FAS had 6MWT done at Week 24, therefore the overall number of participants analyzed is less than the total number of randomized participants.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Molgramostim Once Daily | Molgramostim Intermittent | Placebo
Number analyzed (Participants) | 43 | 43 | 43
meters | 39.6 (95.89) | 11.3 (81.94) | 6.0 (97.17)
Statistical Analysis 1: Comparison: Molgramostim Once Daily vs Placebo; Test type: Superiority; p = 0.3159, ANCOVA; Least Square Means (LSmean) = 20.6, 95% CI 2-sided [-19.8 to 61.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Molgramostim Intermittent vs Placebo; Test type: Superiority; p = 0.7809, ANCOVA; Least Square Means (LSmean) = 5.6, 95% CI 2-sided [-34.1 to 45.2] — [estimate comment as in outcome 1, analysis 2]

3. Secondary Outcome: Change From Baseline in St. George's Respiratory Questionnaire (SGRQ) Total Score After 24 Weeks of Treatment
Description: The SGRQ is designed to measure health impairment in patients with asthma and chronic obstructive pulmonary disease (COPD). It consists of two parts, where Part 1 covers the participants' recollection of their symptoms over the preceding period (1 month recall used in this trial, Symptoms component) and Part 2 addresses the participants' current state in terms of disturbances to their daily physical activity (Activity component) and a wide range of disturbances of psycho-social function (Impact component). A total score as well as individual component scores were calculated. Scores (total and component) range from 0 to 100, with higher scores indicating more limitations.
Time Frame: From baseline to 24 weeks
Population: FAS. Not all participants in the FAS had SGRQ assessed at Week 24, therefore the overall number of participants analyzed is less than the total number of randomized participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Molgramostim Once Daily | Molgramostim Intermittent | Placebo
Number analyzed (Participants) | 45 | 44 | 43
score on a scale | -12.3 (14.30) | -12.0 (15.12) | -4.7 (12.83)
Statistical Analysis 1: Comparison: Molgramostim Once Daily vs Placebo; Test type: Superiority; p = 0.0103, ANCOVA; Least Square Means (LSmean) = -7.6, 95% CI 2-sided [-13.4 to -1.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Molgramostim Intermittent vs Placebo; Test type: Superiority; p = 0.0173, ANCOVA; Least Square Means (LSmean) = -7.0, 95% CI 2-sided [-12.7 to -1.3] — [estimate comment as in outcome 1, analysis 2]

4. Secondary Outcome: Number of Whole Lung Lavage During 24 Weeks of Treatment
Description: In all versions of the protocol (no participants were recruited under version 1.0), whole lung lavage (single lung or both lungs) was applied as rescue therapy. In protocol version 2.0, the criterion for performing whole lung lavage was an increase in (A-a)DO2 by more than 10 mmHg/1.33 kilopascal compared to baseline. In protocol version 3.0 onwards, the criterion for performing whole lung lavage was clinical worsening of aPAP based on symptoms, reduced exercise capacity and/or findings of hypoxemia or desaturation according to the investigator's judgement.
  In protocol versions 2.0 and 3.0, participants undergoing whole lung lavage during the double-blind period were to discontinue double-blind treatment, encouraged to continue to follow the same visit schedule and, if required, receive further whole lung lavage at the investigator's discretion. In protocol version 4.0 and 5.0, participants undergoing whole lung lavage were to continue double-blind treatment.
Time Frame: From baseline to 24 weeks
Population: FAS.
Measure: Number; unit: lavages
Arm/Group | Molgramostim Once Daily | Molgramostim Intermittent | Placebo
Number analyzed (Participants) | 46 | 45 | 47
lavages | 9 | 7 | 17
Statistical Analysis 1: Comparison: Molgramostim Once Daily vs Placebo; Test type: Superiority; p = 0.1918, Negative binomial regression; Risk Ratio (RR) = 0.284, 95% CI 2-sided [0.043 to 1.881] — The estimated value represents the RR between once daily molgramostim and placebo groups
Statistical Analysis 2: Comparison: Molgramostim Intermittent vs Placebo; Test type: Superiority; p = 0.2421, Negative binomial regression; Risk Ratio (RR) = 0.367, 95% CI 2-sided [0.068 to 1.968] — The estimated value represents the RR between intermittent molgramostim and placebo groups

5. Secondary Outcome: Number of Adverse Events (AEs) During 24 Weeks of Treatment
Description: Treatment-emergent adverse events (AEs) were assessed on or after the first dose of trial drug to 28 days after last dose.
  Information about AEs was collected by the investigator by a non-leading question such as "have you experienced any new health problems or worsening of existing conditions" and by reporting events directly observed or spontaneously volunteered by participants (e.g., in the Subject Diary Card, where subjects were asked to record any AEs and answer questions regarding lung toxicity and known systemic effects). Participants were also encouraged to contact the clinic in between visits if they experienced AEs or had any concerns.
  All AEs were assessed by the investigator for severity (mild, moderate, severe), outcome (recovered, not recovered, recovered with sequelae, fatal, unknown) and causality (unlikely, possible, probable, not applicable) according to current regulatory standards.
Time Frame: From baseline to 24 weeks
Population: Safety analysis set: all randomized participants who received at least one dose of the trial drug, analyzed according to actual treatment.
Measure: Number; unit: events
Arm/Group | Molgramostim Once Daily | Molgramostim Intermittent | Placebo
Number analyzed (Participants) | 46 | 45 | 47
events | 215 | 191 | 192

6. Secondary Outcome: Number of Serious Adverse Events (SAEs) During 24 Weeks of Treatment
Description: SAEs are defined as any untoward medicinal occurrence or effect that at any dose:
  * Results in death
  * Is life-threatening
  * Requires hospitalisation or prolongation of existing hospitalisation
  * Results in persistent or significant disability or incapacity
  * Is a congenital anomaly or birth defect
  * May jeopardise the subject or may require intervention to prevent one or more of the other outcomes listed above (Important Medical Events)
Time Frame: From baseline to 24 weeks
Population: Safety analysis set
Measure: Number; unit: events
Arm/Group | Molgramostim Once Daily | Molgramostim Intermittent | Placebo
Number analyzed (Participants) | 46 | 45 | 47
events | 13 | 5 | 16

7. Secondary Outcome: Number of Adverse Drug Reactions (ADRs) During 24 Weeks of Treatment
Description: All AEs judged by either the reporting investigator or the sponsor as having a reasonable causal relationship to a medicinal product qualify as ADRs. The expression reasonable causal relationship means that a causal relationship between a medicinal product and an AE is at least a reasonable possibility i.e. the relationship cannot be ruled out.
Time Frame: From baseline to 24 weeks
Population: Safety analysis set
Measure: Number; unit: events
Arm/Group | Molgramostim Once Daily | Molgramostim Intermittent | Placebo
Number analyzed (Participants) | 46 | 45 | 47
events | 53 | 27 | 33

8. Secondary Outcome: Number of Severe AEs During 24 Weeks of Treatment
Description: All AEs were assessed by the investigator for severity (mild, moderate, severe) according to current regulatory standards:
  * Mild: The AE is easily tolerated and does not interfere with daily activity.
  * Moderate: The AE interferes with daily activity, but the subject is still able to function. Medical intervention may be considered.
  * Severe: The AE is incapacitating and requires medical intervention.
Time Frame: From baseline to 24 weeks
Population: Safety analysis set
Measure: Number; unit: events
Arm/Group | Molgramostim Once Daily | Molgramostim Intermittent | Placebo
Number analyzed (Participants) | 46 | 45 | 47
events | 28 | 11 | 38

9. Secondary Outcome: Number of Participants With at Least 1 AE Leading to Treatment Discontinuation During 24 Weeks of Treatment
Description: Participants could be discontinued from treatment and assessments at any time, if deemed necessary by the investigator. Potential reasons for discontinuation of treatment included e.g. unacceptable AE.
Time Frame: From baseline to 24 weeks
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Molgramostim Once Daily | Molgramostim Intermittent | Placebo
Number analyzed (Participants) | 46 | 45 | 47
Participants | 2 | 1 | 1

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (AEs) were assessed on or after the first dose of trial drug to 28 days after last dose.
Description: Information about AEs was collected by the investigator by a non-leading question such as "have you experienced any new health problems or worsening of existing conditions" and by reporting events directly observed or spontaneously volunteered by participants. Participants were also encouraged to contact the clinic in between visits if they experienced AEs or had any concerns.
Groups:
- Double-blind Molgramostim Intermittent: Inhalation of molgramostim nebuliser solution 300 mcg for 7 days and placebo nebuliser solution for 7 days for 24 weeks (12 cycles)
  Molgramostim: 300 mcg molgramostim (rhGM-CSF) nebulizer solution for inhalation
  Placebo: Placebo nebulizer solution for inhalation
  PARI eFlow nebulizer system: PARI eFlow nebulizer system
Arm/Group | Double-blind Molgramostim Once Daily | Double-blind Molgramostim Intermittent | Double-blind Placebo | Open-label Molgramostim Intermittent
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/45 | 0/47 | 0/130
Serious Adverse Events (participants affected / at risk) | 8/46 | 5/45 | 8/47 | 16/130
Other Adverse Events (participants affected / at risk) | 39/46 | 41/45 | 41/47 | 87/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind Molgramostim Once Daily (N=46) | Double-blind Molgramostim Intermittent (N=45) | Double-blind Placebo (N=47) | Open-label Molgramostim Intermittent (N=130)
Alveolar proteinosis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (3) | 6 (12) | 6 (7)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gambling disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug detoxification (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind Molgramostim Once Daily (N=46) | Double-blind Molgramostim Intermittent (N=45) | Double-blind Placebo (N=47) | Open-label Molgramostim Intermittent (N=130)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (22) | 12 (18) | 11 (12) | 11 (14)
Nasopharyngitis (Infections and infestations) | 7 (10) | 10 (12) | 6 (6) | 24 (33)
Headache (Nervous system disorders) | 6 (9) | 7 (9) | 7 (16) | 3 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (8) | 7 (7) | 4 (5) | 4 (8)
Alveolar proteinosis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 5 (5) | 8 (18) | 7 (10)
Chest pain (General disorders) | 10 (11) | 2 (2) | 1 (2) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (3) | 3 (3) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 6 (6) | 3 (3) | 3 (3)
Pyrexia (General disorders) | 2 (2) | 3 (3) | 3 (4) | 4 (6)
Weight increased (Investigations) | 3 (4) | 5 (6) | 0 (0) | 3 (3)
Respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2) | 2 (2) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3) | 3 (3) | 5 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (5) | 3 (4) | 1 (1) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 4 (4) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2) | 2 (4) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT02702180/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-25): https://cdn.clinicaltrials.gov/large-docs/80/NCT02702180/SAP_001.pdf